CLINICAL TRIAL: NCT05135039
Title: Intervention Effect of Canagliflozin on Prediabetes in Patients With HIV: A Randomized Controlled Trial.
Brief Title: Intervention Effect of Canagliflozin on Prediabetes in Patients With HIV.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: xiaolong zhao (Other)
Responsible Party: Sponsor-Investigator, xiaolong zhao, director, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202140085
Record Dates: First submitted 2021-10-21; First posted 2021-11-26 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: PreDiabetes; Hiv
MeSH Terms: conditions — Prediabetic State; Acquired Immunodeficiency Syndrome | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle interventions + Canagliflozin (Experimental): Subjects were instructed on diet and exercise and advised to make lifestyle changes while they were given daily oral doses of canagliflozin 100mg.
  Interventions: Drug: Canagliflozin
- Lifestyle interventions + Placebo (Placebo Comparator): Subjects were instructed on diet and exercise and advised to make lifestyle changes while they were given daily oral doses of placebo 100mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin 100mg/day/patient
  Arms: Lifestyle interventions + Canagliflozin
Drug: Placebo — Placebo 100mg/day/patient
  Arms: Lifestyle interventions + Placebo

SUMMARY:
The high prevalence of prediabetes in HIV patients is also an outpost event for the further development of diabetes and cardiovascular events, as well as for the prolonged survival of HIV patients with metabolic problems and their complications. Based on the well-established experience in the field of traditional diabetes with prediabetes, the combination of SGLT2 inhibitors can target the pathophysiological mechanisms of HIV-induced metabolic disorders, and the results of a small pilot study of one of the representative drugs, cabergoline, in HIV-combined diabetic patients suggest its efficacy and safety in the treatment of HIV-combined diabetic patients. Combined with the advantages of the concentrated disease resources of HIV patients in the investigator's unit, this study is intended to use a single-center randomized controlled clinical trial design, giving the experimental group drug combined with lifestyle intervention and the control group lifestyle combined with placebo intervention, to verify whether the combination of cabergoline and lifestyle intervention can safely and significantly change the clinical outcome of glucose metabolism, as well as the effect on body weight and pancreatic islet function of patients The study provides top clinical evidence for the treatment of these patients and suggests a new set of interventions for patients with HIV combined with prediabetes. No similar studies have been found to be innovative in the literature search, and the implementation of this study will be of great clinical value.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV infection combined with prediabetes who are not treated with antidiabetic drugs
* Fasting blood glucose of 6.1-6.9 mmol/L or 2-hour oral glucose tolerance test of 7.8-11.0 mmol/L
* BMI >24 kg/m2 and no more than 10% weight fluctuation in 3 months
* HIV-infected patients must be on antiretroviral therapy, no significant symptoms, have HIV RNA below the lower limit of detection for 3 consecutive months, and have CD4 cells greater than 200/uL

Exclusion Criteria:

* Patients with diagnosed diabetes
* Those who are unwilling to participate or unable to cooperate
* The patient has had an acute heart attack or cardiovascular disease in the last three months
* Positive pancreatic islet autoimmune antibody
* History of pancreatitis or pancreatic cancer
* Pregnant or breastfeeding women
* Liver function aminotransferases greater than 2 times the upper limit of the normal range
* Patients with previous recurrent urinary tract infections
* Glomerular filtration rate <45ml/min/1.73m2
* Other serious co-morbidities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of progression from prediabetes to diabetes one year after the intervention in both groups of subjects. | one year
  The rate of progression from prediabetes to diabetes one year after the intervention in both groups of subjects.

SECONDARY OUTCOMES:
Changes in the amount of insulin and C-peptide produced in the two groups of subjects one year after the intervention. | one year
  To investigate the effect of canagliflozin on islet cells, the changes in the amount of insulin and C-peptide produced in two groups of subjects after one year of intervention were examined.
Changes in the number of CD4 T cells after one year intervention in the two groups. | one year
  To investigate whether canagliflozin affects immunity in HIV patients, detect number of CD4T cell changes one year after the intervention in both groups of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Zhao, PhD, Study Chair — Shanghai Public Health Clinical Center
Locations (1):
- Intervention Effect of Canagliflozin on Prediabetes in Patients With HIV: A Randomized Controlled Trial., Shanghai, Shanghai Municipality, China